CLINICAL TRIAL: NCT05795127
Title: Risk for Reoperation After First MTP Joint Arthrodesis
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Mikko Miettinen, M.D., Principal Investigator, Hospital District of Helsinki and Uusimaa
Other Study IDs: HUS/206/2022
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hallux Rigidus; Orthopedic Disorder; Surgery; Complication of Surgical Procedure; Hallux Valgus
Keywords: metatarsal; Hallux rigidus; Hallux valgus
MeSH Terms: conditions — Hallux Rigidus; Musculoskeletal Diseases; Hallux Valgus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reoperated: Primary arthrodesis operations later requiring reoperation.
  Interventions: Procedure: First metatarsophalangeal joint arthrodesis
- Control: Primary arthrodesis operations with no further operations. Size of the control group is four fold.
  Interventions: Procedure: First metatarsophalangeal joint arthrodesis

INTERVENTIONS:
Procedure: First metatarsophalangeal joint arthrodesis — Surgery leadin to bony uninon in firts metatarsophalangeal joint

SUMMARY:
We will screen all first metatarsophalangeal joint arthrodeses performed between 2010 and 2022 in Helsinki University Hospital. Information about demographics and additional diagnoses will be yielded from data pool of medical records. Additionally we review pre- and post-operative x-rays for first MTP joint angles and OR records for operative techniques.

Our aim is to find associations between those known variables and risk for reoperation in two years after operation.

DETAILED DESCRIPTION:
The number of primary surgery in the adult population (age 18 years or older) will be collected from patient information systems using the NOMESCO procedure code NHG80 regardless of diagnosis. These patients will be further screened for diabetes and arthritic diseases (the International Classification of Diseases 10th Revision (ICD-10) diagnostic codes E10.**-E14.** and M05.**-M14.**). As reoperations will be considered surgery under the NOMESCO procedure codes NH***, QDB***, QDG***, ZZH***. Comorbidities were collected from the previous patient health records by diagnosis codes for diabetes type 1 (E10.**), other diabetes (E11.**-14.**), seropositive rheumatoid arthritis (M05.9), seronegative rheumatoid arthritis (M06.0), psoriasis (M07.**), gout (M10.**), other arthritis (M09.**, M11-M14).

The data will be divided and analyzed in two separate phases. First we will gather all the information that we can reliably utilize from the register. The data will include the primary operation, all reoperations, experience level of the surgeon, patients' age, sex, and whether the patient has been diagnosed with other comorbidities stated above.

In the second phase, we will collect matched patients for the patients who underwent reoperations using propensity score matching with ratio of 1:3 with nearest neighbour method. The variables used for matching will be age, sex and all other comorbidities (diabetes type 1, other diabetes, seropositive rheumatoid arthritis, seronegative rheumatoid arthritis, psoriasis, gout, other arthritis) We will further screen the medical records of the reoperated patients as well the matched controls. From pre- and post-operative x-rays we will determine the degree of arthrosis and hallux valgus and intermetatarsal angles. Operation reports will be screened for surgical technique (i.e. method of cartilage removal, fixation and use of bone transport). These data will be used to analyze the association of perioperative factors and reoperations. These models will not be including variables that were used in matching.

During the both phases, we will use logistic regression to analyze association between assumed risk factors and reoperations by using the data from the register (first phase) or from the patients' health records and x-rays (second phase). We will evaluate causality with directed acyclic graphs (DAG), and develop logistic models separately for each of the assumed risk factors. The variables used in the DAGs will be selected based on previous knowledge and hypothesized causal relationships. Results from both analyses will interpreted with adjusted odds ratios (OR) with 95 % confidence intervals (CI). Model fit will be assessed by McFadden R2 -index, multicollinearity by evaluating Variance Inflation Factor (VIF) and heteroscedasticity by inspecting the fitted values vs. residual plots. Statistical analyses will be performed with R version 4.0.5.

ELIGIBILITY:
Inclusion Criteria:

First MTPJ arthrodesis

Exclusion Criteria:

none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated in Helsinki University Hospital in 2010-2022
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of reoperations | 2 years
  Any OR located reoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No